CLINICAL TRIAL: NCT05653128
Title: Food and Nutrition Insecurity During Pregnancy in French Guiana
Acronym: NutriPouTiMoun
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: NutriPouTi'moun
Record Dates: First submitted 2022-11-18; First posted 2022-12-16 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Food Insecurity; Pregnancy Related
Keywords: French Guiana; Pregnancy; Food security; Cross-section study; Nutrition; Social inequality in health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, Hair sample, Cord blood, Placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional study of a representative sample of women who gave birth in the 3 maternity hospitals of French Guiana. The main objective is to estimate the prevalence of food insecurity among pregnant women admitted for delivery in one of the maternity hospitals of French Guiana. A biological assay of deficiencies and toxic metals as well as the completion of a questionnaire will answer the research question

DETAILED DESCRIPTION:
According to the FAO, the gender gap in the prevalence of moderate and severe food insecurity widened in the year of the pandemic, with the prevalence of food insecurity among women 10% higher than among men. Scientific projections have estimated that the increased prevalence of wasting with the pandemic in low- and middle-income countries would result in 18-23% more deaths among children. Worst-case scenarios predict an increase of 8.3 to 38.6% in maternal deaths per month in low- and middle-income countries.

The systemic nature of food insecurity among pregnant women underlines the need to address it in a comprehensive and cross-cutting manner. It seems relevant to consider it as a major determinant of the health of populations that closely follows and feeds other health determinants (precariousness, low standard of living, housing conditions, etc.) or other health consequences (pregnancy monitoring, quality of life, deficiencies, body weight, etc.).

The quality of life would be affected with an increase in stress, anxiety and depression. The link between malnutrition and household food insecurity has already been suggested. Iron deficiency anaemia was significantly associated with food insecurity in the pregnant woman's household; it also predisposes to the risk of anaemia in children under 5. According to the WHO, anaemia is a major public health problem worldwide. It affects 40% of pregnant women, with a risk of irreversible effects on the child's brain development. According to longitudinal studies, the risk of premature delivery seemed to be more frequent when the pregnant woman was in a situation of food insecurity. A diet deficient in essential micronutrients is also thought to increase the risk of low birth weight, according to studies conducted on the African continent.

In Guiana between 2019 and 2020, the CARMA study measured micronutrient deficiencies (Iodine, Iron, Zinc, Vitamin A, folic acid, Vitamin 12) in women at the time of their delivery in Cayenne. This study revealed a high prevalence of micronutrient deficiencies with 81% of parturients having at least 1 deficiency and 46% having at least 2 deficiencies. The authors suggest that the negative impact of heavy metal impregnation is a factor that aggravates deficiencies.

This research takes a global approach to the problem of food security and does not focus on one type of nutritional deficiency or on a pregnancy-related pathology. The idea is to study the links, aggravating effects and interactions between access to food, situations of precariousness, deficiencies, lead or mercury intoxication and the impact with pathologies. This strategy is based on the hypothesis that there are permanent interactions between minerals, vitamins and heavy metals and that their impact on the health of the pregnant woman and the newborn is conditioned by these interactions and by the maternal and family background.

ELIGIBILITY:
Inclusion Criteria:

* Women admitted for delivery in one of the maternity hospitals in French Guiana

Exclusion Criteria:

* refusal to participate or lack of collected non-opposition
* lack of parental consent for women under 18 years of age.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women admitted for delivery in one of the maternity hospitals in French Guiana
Sampling Method: Non-Probability Sample
Enrollment: 788 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Household food insecurity | At inclusion
  The primary measure of household food security was conducted using the Household Food Security Scale (HFSSM) validated by the United States Department of Agriculture (USDA) at inclusion

SECONDARY OUTCOMES:
Evaluation of coping strategies | At inclusion
  Description of the coping strategies using the Coping Strategies Index (CSI) in the past 3 months The Coping Strategy Index (CSI) is an indicator of a household's food security assessing the extent to which households use harmful coping strategies when they do not have enough food or enough money to buy food. The result is reported by a numeric score
Evaluation of the Food Insecurity Experience | At inclusion
  Description of the food insecurity experience using the Food Insecurity Experience Scale (FIES) in the past 3 months The FIES-SM questions refer to the experiences of the individual respondent or of the respondent's household as a whole. The questions focus on self-reported food-related behaviors and experiences associated with increasing difficulties in accessing food due to resource constraints
Evaluation of the food consumption frequencies in the past 3 months | At inclusion
  Description of the food consumption frequencies in the past 3 months using a face-to-face questionnaire
Evaluation of the socio-demographic profile of the household | At inclusion
  Description of the socio-demographic profile of the household at inclusion according to food insecurity level, by face-to-face questionnaire
Evaluation of the economic profile of the household | At inclusion
  Description of the economic profile of the household at inclusion according to food insecurity level, by face-to-face questionnaire
Evaluation of the micronutrient deficiencies | At inclusion
  Evaluation of the micronutrient deficiencies by measuring biomarkers of nutritional status : vitamins and mineral levels, toxic metals in blood and urine
Evaluation of the self esteem | At inclusion
  Description of the self esteem using the Rosenberg Self-Esteem scale by a face-to-face questionnaire The scale ranges from 0-30, with 30 indicating the highest score possible Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Célia BASURKO, MD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (3):
- French Guiana (3):
  - Centre Hospitalier de Cayenne, Cayenne
  - Centre Hospitalier de Kourou, Kourou
  - Centre Hospitalier de l'Ouest Guyanais, Saint-Laurent-du-Maroni

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roberton T, Carter ED, Chou VB, Stegmuller AR, Jackson BD, Tam Y, Sawadogo-Lewis T, Walker N. Early estimates of the indirect effects of the COVID-19 pandemic on maternal and child mortality in low-income and middle-income countries: a modelling study. Lancet Glob Health. 2020 Jul;8(7):e901-e908. doi: 10.1016/S2214-109X(20)30229-1. Epub 2020 May 12. PMID 32405459
- [Background] Pena-Rosas JP, De-Regil LM, Garcia-Casal MN, Dowswell T. Daily oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2015 Jul 22;2015(7):CD004736. doi: 10.1002/14651858.CD004736.pub5. PMID 26198451
- [Background] Aghajafari F, Nagulesapillai T, Ronksley PE, Tough SC, O'Beirne M, Rabi DM. Association between maternal serum 25-hydroxyvitamin D level and pregnancy and neonatal outcomes: systematic review and meta-analysis of observational studies. BMJ. 2013 Mar 26;346:f1169. doi: 10.1136/bmj.f1169. PMID 23533188
- [Background] Hofmeyr GJ, Lawrie TA, Atallah AN, Torloni MR. Calcium supplementation during pregnancy for preventing hypertensive disorders and related problems. Cochrane Database Syst Rev. 2018 Oct 1;10(10):CD001059. doi: 10.1002/14651858.CD001059.pub5. PMID 30277579
- [Background] Wu G, Bazer FW, Cudd TA, Meininger CJ, Spencer TE. Maternal nutrition and fetal development. J Nutr. 2004 Sep;134(9):2169-72. doi: 10.1093/jn/134.9.2169. PMID 15333699
- [Background] Richterman A, Raymonville M, Hossain A, Millien C, Joseph JP, Jerome G, Franke MF, Ivers LC. Food insecurity as a risk factor for preterm birth: a prospective facility-based cohort study in rural Haiti. BMJ Glob Health. 2020 Jul;5(7):e002341. doi: 10.1136/bmjgh-2020-002341. PMID 32611679
- [Background] Moafi F, Kazemi F, Samiei Siboni F, Alimoradi Z. The relationship between food security and quality of life among pregnant women. BMC Pregnancy Childbirth. 2018 Aug 6;18(1):319. doi: 10.1186/s12884-018-1947-2. PMID 30081856
- [Background] Augusto ALP, de Abreu Rodrigues AV, Domingos TB, Salles-Costa R. Household food insecurity associated with gestacional and neonatal outcomes: a systematic review. BMC Pregnancy Childbirth. 2020 Apr 17;20(1):229. doi: 10.1186/s12884-020-02917-9. PMID 32303221
- [Background] Khoshgoo M, Eslami O, Khadem Al-Hosseini M, Shidfar F. The Relationship between Household Food Insecurity and Depressive Symptoms among Pregnant Women: A Cross Sectional Study. Iran J Psychiatry. 2020 Apr;15(2):126-133. PMID 32426008
- [Background] Perez-Escamilla R, Cunningham K, Moran VH. COVID-19 and maternal and child food and nutrition insecurity: a complex syndemic. Matern Child Nutr. 2020 Jul;16(3):e13036. doi: 10.1111/mcn.13036. PMID 32458574
- [Background] Jones AD, Ngure FM, Pelto G, Young SL. What are we assessing when we measure food security? A compendium and review of current metrics. Adv Nutr. 2013 Sep 1;4(5):481-505. doi: 10.3945/an.113.004119. PMID 24038241
- See also: Food security : information for action (practical guides). Introduction to food security concepts — https://www.fao.org/3/al936f/al936f00.pdf
- See also: Summary of World food security status 2021 — https://www.fao.org/3/cb5409fr/cb5409fr.pdf
- See also: Hunger at Covid 19 times in Cayenne (French Guiana) and surroundings — http://beh.santepubliquefrance.fr/beh/2020/29/2020_29_1.html